CLINICAL TRIAL: NCT04369963
Title: The Healthy Endoscopy Study
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Betty Zheng, Principal Investigator, Seattle Children's Hospital
Other Study IDs: STUDY00001638
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Diseases; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Inflammatory Bowel Diseases; Gastrointestinal Diseases | interventions — Endoscopy, Digestive System; Colonoscopy; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — GI tissue biopsies, stool, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Esophagogastroduodenoscopy and Colonoscopy with Biopsies — Participants will have an esophagogastroduodenoscopy and colonoscopy with biopsies. Biopsies from esophagogastroduodenoscopy will not exceed 16 pinch biopsies, biopsies from colonoscopy will not exceed 16 pinch biopsies. Participants will have anesthesia for both procedures.

SUMMARY:
Researchers at Seattle Children's Research Institute want to find ways to understand gastrointestinal disease such as Inflammatory Bowel Disease (IBD), Irritable Bowel Syndrome (IBS) and Graft-Versus-Host-Disease (GVHD). We want to compare healthy cells from the gastrointestinal tract to cells from people with gastrointestinal diseases.

The investigators are looking for healthy participants 18-25 with no gastrointestinal symptoms to volunteer to have an upper and lower endoscopy and to collect blood and stool samples.

The investigators hope the information gathered in this study will help to better predict and treat these diseases in the future.

Participants who join the study will complete the following activities:

1 hour appointment at Seattle Children's Hospital to determine eligibility Blood Draw Upper and Lower Endoscopy with tissue biopsies Stool Sample collection Participants will get $600 to thank them for their time.

Participants may be eligible for this study if they meet the following requirements:

18 -25 years of age Do not have any abdominal symptoms (vomiting, diarrhea or abdominal pain) Are not on any medications (vitamins and birth control are OK) Have a BMI (body mass index) between 20-25 kg/m^2 Please note: Interested participants will have a 30 minute phone call with the study team and subsequent 1 hour appointment at Seattle Children's to determine if they meet all of the eligibility criteria.

DETAILED DESCRIPTION:
This study will enroll a cohort of healthy individuals age 18-25 to volunteer for an esophagogastroduodenoscopy and colonoscopy and will collect of gastrointestinal tissue biopsy samples, blood and stool samples.

Research Procedures include:

* Screening questionnaires
* Medical records review
* Height, weight, blood pressure and temperature measurements
* Collection of urine sample for pregnancy test and banking
* Blood sample up to 50ccs(volume based on weight)
* Stool sample
* GI tissue from endoscopy (4-16 biopsies collected from esophagogastroduodenoscopy, 4 -16 biopsies collected from colonoscopy)

Data to be collected:

* Demographics
* Medical history
* Pregnancy test results
* Endoscopy results
* Pathology results
* Clinical data related to endoscopy
* Clinical lab values

Study population:

The study will enroll 10 participants who meet the following criteria:

* Age 18-25
* No signs or symptoms of present illness
* No known history of chronic illness
* Not on any medications other than birth control or vitamin supplementation
* BMI between 10-25 kg/m^2
* Negative pregnancy test result

Objective/ Purpose:

The samples and information collected from this cohort will be used to understand the mucosal immunity of the gastrointestinal tract in individuals without gastrointestinal problems or history of chronic disease. This information will be used to study the immunology of diseases such as Inflammatory Bowel Disease, Functional Gastrointestinal Disorders and Graft vs. Host Disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -25
* BMI between 20-25
* Participant as no signs or symptoms of present illness
* Participant has no known chronic illness

Exclusion Criteria:

* On medications other than birth control or vitamins
* Pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: You may be eligible for this study if you are:
  18 -25 years of age Do not have any abdominal symptoms (vomiting, diarrhea or abdominal pain) Are not on any medications (vitamins and birth control are OK) Have a BMI (body mas index) between 20-25 Please note: Interested participants will have a 30 minute phone call with the study team and subsequent 1 hour appointment at Seattle Children's to determine if you meet all of the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
To create a single-cell RNA atlas of healthy gastrointestinal tract from healthy participants | 2 years
  A single-cell RNA atlas of the healthy gastrointestinal tract will be created through flow cytometry, T Cell receptor deep sequencing, single cell transcriptome analysis and whole transcriptome analysis on immune cells purified from GI tissue samples and peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Zheng, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Collaborators in Leslie Kean's lab at Boston Children's Hospital will have access to coded data and specimens. Data and specimens that may be shared include: GI tissue samples, whole blood, urine, stool, cDNA, and clinical data without identifying information.
Time Frame: Data and specimens will be stored indefinitely and may be shared at any point in the study's duration
Access Criteria: Study team members at Seattle Children's will have access to patient records and specimens with identification. Collaborator's at Boston Children's will have access to coded specimens and data at request